CLINICAL TRIAL: NCT05901012
Title: Inhaled N,N-Dimethyltryptamine: a Safety and Tolerability Study in Healthy Adults
Brief Title: Safety and Tolerability of DMT in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Draulio Barros de Araujo, PhD, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DMTcog
Record Dates: First submitted 2023-05-22; First posted 2023-06-13 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Safety Issues; Healthy Volunteers
Keywords: N,N-DMT; N,N-Dimethyltryptamine; DMT; placebo; psychedelic
MeSH Terms: interventions — N,N-Dimethyltryptamine

STUDY DESIGN:
Intervention Model Description: This is a double-blind, randomized, placebo-controlled crossover design. 25 participants will be evaluated, who will undergo two dosing sessions on the same day: with DMT (60 mg, inhaled) and with placebo (1 mg DMT, inhaled). Each session will last approximately 2 hours, the substance order will be randomized.
Who Masked: Participant, Investigator
Masking Description: This study employs a double-blind design. The participant and investigator will all be blind to the order of substance administration during the dosing sessions. Each participant will undergo two dosing sessions on the same day, one with N,N-Dimethyltryptamine (DMT) at a dosage of 60 mg, and another with a placebo containing 1 mg of DMT. The order of substance administration (DMT or placebo) will be randomized and unknown to all parties involved in the study until data collection is complete to ensure unbiased results
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 60mg of N,N-Dimethyltryptamine (Experimental): One inhaled dose of 60mg of vaporized DMT.
  Interventions: Drug: N,N-Dimethyltryptamine
- Placebo-like (Placebo Comparator): One inhaled dose of 1mg of vaporized DMT.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N,N-Dimethyltryptamine — DMT will be administered using a vaporizer device in a placebo-controlled, double-blind, randomized, monocentric clinical trial design.
  Other Names: DMT
  Arms: 60mg of N,N-Dimethyltryptamine
Drug: Placebo — DMT will be administered using a vaporizer device in a placebo-controlled, double-blind, randomized, monocentric clinical trial design.
  Arms: Placebo-like

SUMMARY:
This study aims to evaluate the acute and subacute effects of an inhaled N, N-Dimethyltryptamine (DMT) in healthy individuals.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled crossover design. 25 participants will be evaluated, who will undergo two dosing sessions on the same day: with DMT (60 mg, inhaled) and with placebo (1 mg DMT, inhaled). Each session will last approximately 2 hours; the substance order will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* previous experience with DMT
* be right-handed
* healthy volunteers

Exclusion Criteria:

* heart failure
* liver failure
* kidney failure
* uncontrolled high blood pressure
* history of heart rhythm disorders
* history of valvular heart disease
* history of chronic obstructive pulmonary disease (COPD)
* active or in treatment for bronchial asthma
* severe obesity
* coagulation disorders
* clinical evidence or history of increased intracranial
* clinical evidence or history of cerebrospinal pressure
* history or reports of epilepsy
* severe neurological disease,
* pregnancy
* reported or clinically recognized thyroid disorders
* diagnosis or family suspicion of genetic monoamine deficiency oxidase
* previous adverse response to psychedelic substances
* symptoms or family members with a present or past psychotic disorder
* dissociative identity disorder
* bipolar affective disorder
* prodromal symptoms of schizophrenia
* problematic use or abuse of alcohol or other psychoactive substances (except tobacco)
* acute or subacute risk of suicide
* acute flu symptoms
* symptoms of airway infection
* contact with a confirmed case of COVID-19 (SARS-CoV-2) in the last 7 days

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-17 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure | up to 2 hours
  Assessed 7 times on each session
Diastolic Blood Pressure | up to 2 hours
  Assessed 7 times on each session
Heart rate | up to 2 hours
  Assessed 7 times on each session
Respiratory rate | up to 2 hours
  Assessed 7 times on each session
Oxygen saturation | up to 2 hours
  Assessed 7 times on each session

SECONDARY OUTCOMES:
Plasma level of glucose | up to 2 hours
  Assessed 2 times on each session
Plasma level of total cholesterol | up to 2 hours
  Assessed 2 times on each session
Plasma level of C-reactive protein (CRP) | up to 2 hours
  Assessed 2 times on each session
Plasma level of urea | up to 2 hours
  Assessed 2 times on each session
Plasma level of creatinine | up to 2 hours
  Assessed 2 times on each session
Plasma level of aspartate transaminase (AST) | up to 2 hours
  Assessed 2 times on each session
Plasma level of alanine transaminase (ALT) | up to 2 hours
  Assessed 2 times on each session
Plasma level of cortisol | up to 2 hours
  Assessed 2 times on each session
Plasma level of subjective effects of DMT | up to 2 hours
  Assessed 2 times on each session
Evaluate the subjective effects of DMT | up to 2 hours
  Assessment of the acute subjective effects of DMT, compared to placebo, by 5D-ASC (5 Dimensions- Altered States of consciousness). Scores range from 0 to 94, where higher scores indicate more intense psychedelic subjective effects.
Evaluate the subjective effects of DMT | up to 2 hours
  Assessment of the acute subjective effects of DMT, compared to placebo, by HRS (Hallucinogen Rating Scale). Scores range from 0 to 400, where higher scores indicate more intense psychedelic subjective effects.
Evaluate the subjective effects of DMT | up to 2 hours
  Assessment of the acute subjective effects of DMT, compared to placebo, by MEQ (Questionnaire of Mystical Experiences). Scores range from 0 to 150, where higher scores indicate more intense psychedelic subjective effects.
Evaluate acute effects on alpha waves using electroencephalography before, during and after the dosing | up to 1 hours
  Assessment of the electrical cerebral activity in different bandwidth as alpha waves by EEG before, during and after each session.
Evaluate acute effects on beta waves using electroencephalography before, during and after the dosing | up to 1 hours
  Assessment of the electrical cerebral activity in different bandwidth as beta waves by EEG before, during and after each session.
Evaluate acute effects on theta waves using electroencephalography before, during and after the dosing | up to 1 hours
  Assessment of the electrical cerebral activity in different bandwidth as theta waves by EEG before, during and after each session.
Evaluate the subacute effects of DMT, compared to placebo, on electroencephalography markers | up to 0.5 hours
  Assessment of the subacute effects of DMT on EEG, including ERP (event-related potential ) generated from visual and auditory stimulation by applying a visual and auditory perception and imagination task.
Evaluate the acute effects of DMT, compared to placebo, on electroencephalography markers | up to 0.5 hours
  Assessment of the acute effects of DMT in ERP (event-related potential) generated from auditory stimulation in an oddball protocol.
Evaluate the subacute effects of DMT on suggestibility | up to 1 hours
  Assessment of the subacute effects of DMT on suggestibility by applying a suggestibility task named Creative Imagination Scale (CIS). Scores range from 0 to 40. Higher scores indicate more intense suggestibility.
Evaluate the influence of expectations | up to 0.5 hours
  Assessment of the influence of expectations variables on subjective experience
Evaluate the influence of personality trait | up to 0.5 hours
  Assessment of the influence of personality trait on suggestibility
Assess DMT Plasma Concentration-Time Profile using High-performance liquid chromatography | up to 50 minutes
  Evaluate changes in serum DMT concentration over time measured in baseline, 2 and 50 minutes after each session.

CONTACTS AND LOCATIONS:
Overall Officials: Draulio B. Araujo, Ph.D, Principal Investigator — Universidade Federal do Rio Grande do Norte
Locations (1):
- Hospital Universitário Onofre Lopes, Natal, Rio Grande do Norte, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wiessner I, Falchi-Carvalho M, Laborde S, Barros H, Bolcont R, Ruschi Silva S, Pantrigo E, Medina M, Arichelle F, Almeida R, Aires R, Nunes Ferreira LF, Dantas Correa L, Da Costa Bezerra RB, Thie K, Silva-Costa N, de Araujo Costa Neto LA, Jales Lima de Queiroz MV, Galvao-Coelho N, Araujo D, Palhano-Fontes F. Safety, tolerability and subjective effects of vaporized N,N-Dimethyltryptamine: A randomized double-blind clinical trial. Eur Neuropsychopharmacol. 2025 Aug;97:16-27. doi: 10.1016/j.euroneuro.2025.06.002. Epub 2025 Jun 17. PMID 40532423
- See also: Hospital Universitário Onofre Lopes - UFRN (Federal University of Rio Grande do Norte) — https://www.gov.br/ebserh/pt-br/hospitais-universitarios/regiao-nordeste/huol-ufrn